CLINICAL TRIAL: NCT02312518
Title: A Prospective, Randomized Clinical Trial of PRP Concepts Fibrin Bio-Matrix in Chronic Non-Healing Venous Leg Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PRP Concepts, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PC003
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Venous Leg Ulcers
Keywords: non-healing wounds; venous stasis; ulcer; platelet rich plasma
MeSH Terms: conditions — Varicose Ulcer; Ulcer | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- PRP Concepts Fibrin Bio-Matrix (Experimental): PRP Concepts Fibrin Bio-Matrix in addition to usual and customary practice
  Interventions: Device: PRP Concepts Fibrin Bio-Matrix; Other: Usual and Customary Practice
- Usual and Customary Practice (Other): usual and customary practice
  Interventions: Other: Usual and Customary Practice

INTERVENTIONS:
Device: PRP Concepts Fibrin Bio-Matrix — PRP Concepts Fibrin Bio-Matrix in addition to usual and customary practice
  Arms: PRP Concepts Fibrin Bio-Matrix
Other: Usual and Customary Practice — Usual and Customary Practice for non-healing venous leg ulcers
  Other Names: Standard of Care

SUMMARY:
To assess the efficacy of the PRP Concepts Fibrin Bio-Matrix and compare its performance with usual and customary practice for the treatment of chronic non-healing venous leg ulcers (VLU).

DETAILED DESCRIPTION:
This is a prospective, randomized, single-blind, controlled, multi-center study for subjects undergoing VLU treatment. Qualified subjects will be randomized (1:1); test group (PRP Concepts Fibrin Bio-Matrix) and control group (usual and customary practice). The study will consist of 3 periods: a screening period, an active treatment period, and a follow-up period (if healed). Approximately 250 subjects will be enrolled. Subjects will be ≥18 years of age with a VLU (greater than 4 weeks duration). Each subject will be enrolled in the active treatment period for up to 12 weeks, or to closure of wound with a confirmatory visit 2 weeks after wound closure, whether such closure occurs at 12 weeks or earlier.

ELIGIBILITY:
Inclusion Criteria:

Medicare/Medicaid eligible Proven venous disease The index ulcer is greater than 4 weeks duration. Three or fewer ulcers that are separated by > 3.0 cm distance The largest non-healing wound, if multiple wounds are present, or the single wound to be treated (Index Ulcer) that is located between and including the knee and the ankle Post-debridement, the ulcer size must be between 2 cm2 and 200 cm2 Demonstrated adequate compression regimen Able and willing to attend scheduled follow-up visits and study related exams Able and willing to provide a voluntary written informed consent.

Exclusion Criteria:

Ulcer not of VLU pathophysiology (e.g., pure diabetic, vasculitic, radiation, rheumatoid, collagen vascular disease, pressure, or arterial etiology) Greater than 30% reduction in wound size during the first two weeks of observation and treatment by the investigator Gross clinical infection at the study ulcer site including cellulitis and osteomyelitis. Known allergy tor sensitivity to Eclipse PRP kit components (calcium chloride, calcium gluconate or acid citrate dextrose solution A (ACDA)) Serum albumin of less than 2.5 g/dL, Plasma Platelet count of less than 100 x 109/L, or Hemoglobin of less than 10.5 g/dL, Known renal failure as determined by a Creatinine > 2.5 mg/dl Malignancy at or near the ulcer site Rheumatoid arthritis (and other collagen vascular disease), vasculitis, sickle cell disease, HIV Severe liver disease. Presence of additional abnormal lab values obtained within 7 days prior to the Day 0 visit determined to be clinically significant by the investigator including: WBC >13,000/cm3 or < 5, 000 cm3, or electrolytes that are outside the host institution's range of normal Radiation therapy, chemotherapy, immunosuppressive therapy or chronic steroid use within 30 days of enrollment Received another investigational device or drug within 30 days of enrollment Received allograft, autograft or xenograft within 30 days of enrollment Subject has inadequate venous access for repeated blood draw required for Eclipse RPR administrations Subject requires or is anticipated to require interventions directed at improvement of arterial perfusion to affected area Ulcer expected to be treated with any advanced therapeutics (e.g., HBOT) Presence of another wound that is concurrently treated and might interfere with treatment of index wound Subjects who are cognitively impaired and do not have a healthcare proxy Life expectancy of < 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to complete wound closure | 12 weeks
  Complete wound closure is defined as full epithelialization of the wound with the absence of drainage, durability confirmed at 2 weeks
Percent of wounds healed | 12 weeks
  Percent of wounds healed at 12 weeks

SECONDARY OUTCOMES:
Wound Trajectory | 12 weeks
  Mean and median of percent (%) wound size changes at 4 weeks, 8 weeks and 12 weeks
Ulcer recurrence | 3 months
  Ulcer recurrence out to 3 months for subjects whose wounds heal by conclusion of 12 weeks visit.
Quality of Life Health Survey | 3 months
  Changes in Quality of Life scores and ability to return to previous function/resumption of normal activities

CONTACTS AND LOCATIONS:
Overall Officials: Damon Keeley, Study Director — PRP Concepts, LLC
Locations (1):
- Westchester General Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No